CLINICAL TRIAL: NCT05876182
Title: A Prospective, Randomized, Placebo-controlled Clinical Trial of Oral Vancomycin in Adults and Young Adults (15-17 Years Old) Affected by Primary Sclerosing Cholangitis With or Without Inflammatory Bowel Disease
Brief Title: Vancomycin in Primary Sclerosing Cholangitis in Italy
Acronym: VanC-IT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Collaborators: Genetic s.p.a. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VanC-IT
Record Dates: First submitted 2023-03-10; First posted 2023-05-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Primary Sclerosing Cholangitis; Liver and Intrahepatic Bile Duct Disorder; IBD
Keywords: liver; oral vancomycin; primary sclerosing cholangitis; Inflammatory bowel disease
MeSH Terms: conditions — Cholangitis, Sclerosing; Digestive System Diseases; Inflammatory Bowel Diseases | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: Group A: vancomycin 750 mg daily Group B: vancomycin1500mg daily Group C: placebo
Who Masked: Participant, Investigator
Masking Description: During the randomization phase, subjects and all personnel directly involved in the conduct of the study will be blinded to the treatment assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Vancomycin 750 (Experimental): 28 subjects with PSC will be randomized to this arm. They will take 2 tablet (1 of vancomycin 250 mg and 1 of placebo), three times a day administered orally (total dose 750 mg/daily).
  Interventions: Drug: Oral Vancomycin
- Oral Vancomycin 1500 (Experimental): 28 subjects with PSC will be randomized to this arm.They will take 2 tablet of 250 mg of vancomycin three times a day administered orally (total dose 1500mg/daily)
  Interventions: Drug: Oral Vancomycin
- Placebo (Placebo Comparator): 28 subjects with PSC will be randomized to this arm. They will take 2 tablet (placebo-to-match oral vancomycin) administered orally three times a day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oral Vancomycin — The investigator will identify potential participants and confirm the diagnosis of PSC. Subjects will be screened within 10 weeks before randomization to determine the eligibility. Study participants will be consecutively randomized to oral vancomycin or placebo and investigational drug and placebo dispensed.
  Other Names: OV
  Arms: Oral Vancomycin 1500; Oral Vancomycin 750
Other: Placebo — The investigator will identify potential participants and confirm the diagnosis of PSC. Subjects will be screened within 10 weeks before randomization to determine the eligibility. Study participants will be consecutively randomized to oral vancomycin or placebo and investigational drug and placebo dispensed.
  Arms: Placebo

SUMMARY:
Primary sclerosing cholangitis (PSC) is chronic fibroinflammatory disease of the liver. There is still no medical therapy proven to halt the progression of PSC or prevent its serious complications.

This is a Phase 2 randomized, double bind, placebo-controlled, monocentric study evaluating the safety and efficacy of two doses of oral vancomycin (i.e. 750 mg and 1500 mg/day) in subject between 15 - 70 years old with PSC.

DETAILED DESCRIPTION:
Primary sclerosing cholangitis (PSC) is chronic fibroinflammatory disease of the liver characterized by chronic inflammation and sclerosis of the intrahepatic and/or extrahepatic bile ducts, and a risk for progression to liver failure and development of colorectal and hepatobiliary cancer. Both children and adults are affected. Patients with PSC have a diminished life expectancy with a median survival of 17 years after diagnosis. Despite the high mortality associated with PSC and the efforts to optimize its management, there is no medical therapy proven to halt the progression of PSC or prevent its serious complications. There is a strong yet poorly understood relationship between PSC and inflammatory bowel disease (IBD); nearly 70%-80% of PSC patients have IBD, mainly ulcerative colitis (UC). Increasing evidence is pointing out the role of gut microbiota in the pathogenesis of PSC. The 'leaky gut' theory implies that either bacteria or their toxic metabolites translocate from the inflamed intestinal mucosa into the portal circulation and into the liver causing liver and biliary injury. The gut microbiota of PSC patients, compared to IBD patients and healthy controls, showed decreased microbial diversity, and over-represented intestinal pathobionts (i.e., organisms which, under normal circumstances, lives as a non-harming symbiont). Several antibiotics, including vancomycin and metronidazole, have been investigated in PSC. The use of oral vancomycin (OV), a glycopeptide antibiotic has been reported to be associated with improvement in clinical symptoms and laboratory abnormalities in patients with PSC; however, prospective studies in adult and young adult patients in Europe are lacking.

Our scientific community therefore seeks to examine the safety and efficacy of OV in patients with PSC in a randomized placebo-controlled clinical trial.

This is a Phase 2 randomized, double bind, placebo-controlled, monocentric study evaluating the safety and efficacy of two doses of oral vancomycin (i.e. 750 mg and 1500 mg/day) in subject between 15 - 70 years old with PSC with or without IBD. The study will consist of 10-week screening period (including a run-in phase), 24 weeks of treatment, and follow-up visits at 4 and 12 weeks after completion of treatment to evaluate what happens after treatment stop. Subjects will be randomized to placebo or treatment and stratifying by baseline presence of fibrosis by fibroscan value at baseline (< or ≥14.4 kPa corresponding to F4 fibrosis), as this parameter could affect the likelihood of reaching the primary composite outcome measure.

The knowledge gained from our proposed clinical trial will help us determine if OV should be considered as a treatment option in patients with PSC. Furthermore, the use of state-of-the art technology applied in this study will shed light on the relationship between the gut microbiome, bile acids, immune-mediators, including cytokines, and PSC.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give informed consent prior to any study specific procedure being performed;
2. Male and non-pregnant, non-lactating female subjects, including women of child bearing potential (WOCBP), between 15-70 years of age at the time of informed consent;
3. Diagnosis of large-duct PSC based on cholangiogram (at MRCP, ERCP, PTC) according to the most recent published guidelines (EASL);
4. Baseline ALP ≥1.5 times upper limit normal at screening;
5. Absence of biliary obstruction and/or malignancy within 6-12 months of entry into the study;
6. If a patient is on ursodeoxycholic acid (UDCA) or 5-aminosalicylic acid he or she is expected to remain on the same daily dose during the study period;
7. Patients who received antibiotics or probiotics may participate if they had a washout period of at least 3-month prior to study entry;
8. If a patient has been on obeticholic acid or other experimental therapies (e.g. cilofexor and norUDCA) for PSC, they must complete a 3-month washout period before study entry;
9. PSC with or without IBD. IBD diagnosis should be documented and with a minimum disease duration of 6 months, as determined by endoscopic and histopathology assessment. IBD should be in clinical remission or mildly active according to CDAI and partial Mayo score for CD and UC, respectively (i.e. patients with CDAI score < 220 and pMayo score <5). Patients without documented IBD need a colonoscopy with segmental biopsies within 12 months prior to baseline visit;
10. Female subjects of childbearing potential must test negative for pregnancy at screening, baseline and follow-up visits and if engage in sexual intercourse must agree to use specific methods of contraception.
11. Male subjects with female partners of childbearing potential must use condoms during treatment and until the end of relevant systemic exposure.

Exclusion Criteria:

1. Receiving an antibiotic or probiotic within 3 months prior to the study;
2. Expected to receive antibiotics within the weeks leading up to enrollment (such as patients with recurrent cholangitis, ongoing infectious illnesses, etc.);
3. Allergy to vancomycin or teicoplanin;
4. Biliary intervention within 3 months prior to study enrollment or planned;
5. Alcohol abuse (defined as greater than 14 standard drinks units per week in men; greater than 7 standard drinks units per week);
6. Pregnancy and lactation;
7. Advanced renal disease (GFR< 70);
8. Active hepatitis B and/or C infection;
9. Other chronic or cholestatic liver diseases such as PBC, autoimmune hepatitis, nonalcoholic steatohepatitis, alcoholic liver disease, Wilson's disease, hemochromatosis, α-1 antitrypsin deficiency, IgG4-related sclerosing cholangitis, and liver cancer;
10. History of CCA;
11. Advanced liver disease (history of variceal bleeding, ascites, hepatic encephalopathy, and/or bilirubine >4 mg/dL);
12. On active transplantation list;
13. IBD with uncontrolled moderate to severe activity;
14. Active treatment or within the previous four weeks (washout period) with any immunosuppressive medication for controlling IBD (i.e. azathioprine, 6-mercaptopurine, tacrolimus, methotrexate, infliximab, adalimumab, golimumab, vedolizumab, ustekinumab, tofacitinib, ozanimod). Treatment with corticosteroids (including budesonide, budesonide MMX and beclomethasone) in the previous four weeks
15. Active treatment with rifampicin or within the previous three months (washout period);
16. Dose change within last 3 months prior to baseline of concomitant treatment with vitamin D or fibrates;
17. Treatment with any experimental drug within the previous three months;
18. Any known relevant infectious disease (e.g. active tuberculosis, AIDS defining disease);
19. History or active hearing problems;
20. Any active malignant disease;
21. Well found doubt about patient's cooperation, e.g. addiction to alcohol or drugs;
22. Imprisoned person, person admitted to nursing homes, persons under legal guardianship, and persons not able to express their consent.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in alkaline phosphatase (ALP) levels | From baseline to 6 months
  ALP levels at 6 months

SECONDARY OUTCOMES:
Safety and tolerability of OV in each treatment arm | From baseline to 6 months
  Adverse events
Clinical hematology | From baseline to 6 months
  White blood cells (10^3/uL)
Clinical hematology | From baseline to 6 months
  Hemoglobin (g/dl)
Clinical hematology | From baseline to 6 months
  Hematocrit (%)
Clinical hematology | From baseline to 6 months
  MCV (Mean Corpuscular Volume) (fL)
Clinical hematology | From baseline to 6 months
  Platelets (10^3/uL)
Clinical hematology | From baseline to 6 months
  Absolute neutrophils (10^3/uL)
Clinical hematology | From baseline to 6 months
  Absolute lymphocytes (10^3/uL)
Clinical hematology | From baseline to 6 months
  PT (Prothrombin Time, Ratio)
Clinical hematology | From baseline to 6 months
  INR
Clinical chemistry | From baseline to 6 months
  Total proteins (g/dl)
Clinical chemistry | From baseline to 6 months
  Albumin (g/dl)
Clinical chemistry | From baseline to 6 months
  Gamma (g/dl)
Clinical chemistry | From baseline to 6 months
  Sodium (mmol/l)
Clinical chemistry | From baseline to 6 months
  Creatinine (mg/dl)
Clinical chemistry | From baseline to 6 months
  Potassium (mmol/l)
Clinical chemistry | From baseline to 6 months
  Urea (mg/dl)
Clinical chemistry | From baseline to 6 months
  Glucose (mg/dl)
Clinical chemistry | From baseline to 6 months
  Total bilirubin (mg/dl)
Clinical chemistry | From baseline to 6 months
  Direct bilirubin (mg/dl)
Clinical chemistry | From baseline to 6 months
  GGT (U/l)
Clinical chemistry | From baseline to 6 months
  AST (U/l)
Clinical chemistry | From baseline to 6 months
  ALT (U/l)
Clinical chemistry | From baseline to 6 months
  Triglycerides (mg/dl)
Clinical chemistry | From baseline to 6 months
  Cholesterol (Total) (mg/dl)
Clinical chemistry | From baseline to 6 months
  High Density Lipoprotein (HDL Cholesterol) (mg/dl)
Clinical chemistry | From baseline to 6 months
  PCR (C Reactive Protein) (mg/dl)
Clinical chemistry | From baseline to 6 months
  IgG (mg/dl)
Clinical chemistry | From baseline to 6 months
  IgA (mg/dl)
Clinical chemistry | From baseline to 6 months
  IgM (mg/dl)
Clinical chemistry | From baseline to 6 months
  Ferritin (ng/ml)
Single 12-lead electrocardiograms | From baseline to 6 months
  Sinus rhythm
Single 12-lead electrocardiograms | From baseline to 6 months
  QTc (msec)
Urine analysis | From baseline to 6 months
  pH
Urine analysis | From baseline to 6 months
  Specific gravity
Urine analysis | From baseline to 6 months
  Hemoglobin
Urine analysis | From baseline to 6 months
  ACR (mg/g)
Urine analysis | From baseline to 6 months
  PCR (mg/g)
Vital sign measurements | From baseline to 6 months
  Body weight (kg)
Vital sign measurements | From baseline to 6 months
  Systolic blood pressure (mmHg)
Vital sign measurements | From baseline to 6 months
  Diastolic blood pressure (mmHg)
Vital sign measurements | From baseline to 6 months
  Heart Rate (bpm)
Vital sign measurements | From baseline to 6 months
  Temperature (°C)
Changes in the PSC score | From baseline to 6 months
  Revised Mayo Risk Score (Calculation formula = 0.03 (age [y]) + 0.54 loge (bilirubin [mg/dL]) + 0.54 loge (aspartate aminotransferase [U/L]) + 1.24 (variceal bleeding [0/1]) - 0.84 (albumin [g/dL]) (Higher scores indicate greater disease severity)
Changes in the IBD score | From baseline to 6 months
  Clinical Mayo Score (Partial Mayo Score) -(0-1=Remission; 2-4 = Mild activity; 5-7 = Moderate activity; 7-9 = Severe activity)
Liver stiffness measurements | From baseline to 6 months
  Stiffness (kPa/s)
Liver stiffness measurements | From baseline to 6 months
  Stiffness IQR/median (%)
Liver stiffness measurements | From baseline to 6 months
  CAP (dB/m)
Liver stiffness measurements | From baseline to 6 months
  CAP IQR/median (%)
MRCP (Magnetic Resonance Cholangiopancreatography) | From baseline to 6 months
  Disease localisation
MRCP (Magnetic Resonance Cholangiopancreatography) | From baseline to 6 months
  Presence of dominant stenosis
MRCP (Magnetic Resonance Cholangiopancreatography) | From baseline to 6 months
  Radiological signs of cirrhosis
Cytokines changes | From baseline to 6 months
  TGF-β levels
Cytokines changes | From baseline to 6 months
  IL-4 levels
Cytokines changes | From baseline to 6 months
  IL-13 levels
Cytokines changes | From baseline to 6 months
  IL-10 levels
Changes in the peripheral blood mononuclear cells | From baseline to 6 months
  Th1 and Th17 subsets isolation and analyses
Patients quality of life | From baseline to 6 months
  Visual analogue scale (VAS) score for itch
Patients quality of life | From baseline to 6 months
  Chronic Liver Disease Questionnaire (CLDQ)
Patients quality of life | From baseline to 6 months
  EQ-5D-5L questionnaire
Patients quality of life | From baseline to 6 months
  PSC patient reported outcome (PSC-PRO) questionnaire
Patients quality of life | From baseline to 6 months
  Inflammatory Bowel Disease Questionnaire (IBDQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza E Brianza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cristoferi L, D'Amato D, Maino C, Bernasconi D, Dinelli ME, Malandrin SMI, Facciotti F, Festa MM, Gerussi A, Rossi E, Malinverno F, Tettamanti P, Cazzaniga ME, Corso R, Ippolito D, Galimberti S, Invernizzi P, Carbone M. Prospective, randomised, placebo-controlled, phase 2 clinical trial assessing the efficacy and safety of oral vancomycin in patients with primary sclerosing cholangitis with/out inflammatory bowel disease in Italy: study protocol of VanC-IT trial. BMJ Open. 2026 Jan 9;16(1):e106630. doi: 10.1136/bmjopen-2025-106630. PMID 41513411